CLINICAL TRIAL: NCT01028612
Title: A Pilot Study of Interventional Thermal Ablation Combined With External Beam Radiation Therapy for Patients With Inoperable Non-Small Cell Lung Cancer > 3.5 cm in Size
Brief Title: Thermal Ablation Combined With External Beam Radiation Therapy for Patients With Inoperable Non-Small Cell Lung Cancer > 3.5 cm in Size
Acronym: NSCLC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011975; CCCWFU 62109 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- thermal ablation with external beam radiation (Experimental)
  Interventions: Radiation: thermal ablation with external beam radiation

INTERVENTIONS:
Radiation: thermal ablation with external beam radiation — thermal ablation with external beam radiation

SUMMARY:
The main objective of this study is to assess the initial safety of the combination of interventional ablation and external beam radiotherapy including acute and late toxicity (90 days) for patients with early stage lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AJCC sixth edition Stage Ib or II non-small-cell lung cancer with cytology or biopsy proven disease and a minimum tumor size of 3.5 cm are eligible.
* To be considered node negative for N2 disease, patients will have mediastinal lymph nodes ≤ 1.5 cm and no clinically suspicious uptake on FDG PET in those areas.
* All patients are required to have been evaluated by a thoracic surgeon and have either refused surgery or been deemed medically inoperable due to co-morbid conditions.
* The CT images of the chest must be reviewed by an experienced interventional radiologist and the target lesion is determined to be in a location where RFA is technically achievable based on the proximity of adjacent organs and structures.
* Age ≥ 18 years old
* Performance Status 0-2 (ECOG)

Exclusion Criteria:

* History of prior malignancy within the past 2 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, T1N0 squamous cell carcinoma of the larynx, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry
* Previous chest radiation to the region of interest.
* Pregnant or lactating women.
* A clinical diagnosis of bronchoalveolar carcinoma (BAC) will be made for patients in whom tissue diagnosis is by cytology alone with adenocarcinoma shown and the following radiographic criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Assess the initial safety of the combination of interventional ablation and external beam radiotherapy including acute and late toxicity (90 days). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States